CLINICAL TRIAL: NCT01303575
Title: It's Your Game...Keep It Real for American Indian/Alaska Native Youth: Innovative Approaches to Prevent Teen Pregnancy Among Underserved Populations
Brief Title: Internet-Based Sexual Health Education for Middle School Native American Youth
Acronym: IYG-AI/AN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Alaska Native Tribal Health Consortium (Other); Inter Tribal Council of Arizona (Unknown); Northwest Portland Area Indian Health Board (Other)
Responsible Party: Principal Investigator, Ross Shegog, Associate Professor - School of Public Health, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 5U48DP001949 (NIH)
Record Dates: First submitted 2011-02-18; First posted 2011-02-24 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2013-11

CONDITIONS: Sexually Transmitted Diseases; Pregnancy; HIV Infections
Keywords: Adolescents; Youth; Sexual Health; Sex Education; Pregnancy Prevention; Abstinence Education; HIV; Human Immunodeficiency Virus; STI; Chlamydia; Gonorrhea; Sexually Transmitted Infections; American Indian; Alaska Native; Native American; Internet-Based; Computer-based Education; Computer-based learning
MeSH Terms: conditions — Sexually Transmitted Diseases; HIV Infections; Acquired Immunodeficiency Syndrome; Chlamydia Infections; Gonorrhea | interventions — Seroconversion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HIV, STI, and Pregnancy Prevention Curriculum (Experimental)
  Interventions: Behavioral: HIV, STI and Pregnancy Prevention Curriculum
- Control curricula: Science Education (Active Comparator): No sexual health elements
  Interventions: Behavioral: Control Curricula

INTERVENTIONS:
Behavioral: HIV, STI and Pregnancy Prevention Curriculum — A complete internet-based, "It's Your Game...Keep It Real" Intervention Program
  Arms: HIV, STI, and Pregnancy Prevention Curriculum
Behavioral: Control Curricula — A computer-based, science education program that does not contain elements of sexual health education
  Arms: Control curricula: Science Education

SUMMARY:
This study will evaluate the effect of an American Indian/Alaska Native (AI/AN) adaptation of the It's Your Game…Keep It Real (IYG) intervention, relative to a comparison condition on sexual behavior outcomes and psychosocial variables for middle school aged youth (12 - 14 years old). The original IYG program was designed for students in Houston middle schools to help students delay sexual initiation and if sexually active, use condoms and contraception. The present study will adapt the existing IYG program for an AI/AN youth cohort; the original IYG curriculum will be transferred into a web-based format and modified to incorporate additional culturally-relevant components. The primary hypothesis to be tested is: (1) students who receive the web-based curriculum will delay sexual activity relative to those who receive standard care. The major dependent variable is the proportion of students initiating sexual activity. Secondary hypotheses will examine the effect of the web-based curriculum on specific types of sex and psychosocial variables related to sexual risk-taking behavior. This project will also examine the effect of the intervention on the proportion of students who are sexually active, number of times students engage in unprotected sexual intercourse, and students' number of sexual partners.

DETAILED DESCRIPTION:
The goal of this four year research project is to adapt and evaluate the effectiveness of an Internet-based HIV/STI, and pregnancy prevention curriculum for American Indian/Alaska Native (AI/AN) middle school-aged youth (12-14 years). This curriculum will be adapted from a successful, Internet-accessible, prevention program, It's Your Game…Keep it Real (IYG).

During year 1 (Fall 2010 through Spring 2011) of this project, the study team will test the usability of the existing IYG program, while performing an assessment of existing programs for cultural of the IYG intervention. In year 2 (beginning Fall 2011), the project team plans to initiate and complete development of the cultural-adapted IYG intervention for AI/AN youth (IYG-AI/AN). Starting in year 3 (Fall 2012), the study efficacy trial will commence to evaluate the effectiveness of IYG-AI/AN on sexual behaviors and psychosocial determinants of those behaviors among AI/AN youth in three regions (Alaska, the Pacific Northwest, including Idaho, Oregon, and Washington state, and Arizona) relative to a comparison condition. Recruitment sites will be middle schools and Boys and Girls Clubs (BGCs), identified through their affiliations with the Alaska Native Tribal Health Consortium (ANTHC), the Pacific Northwest Tribal Epicenter (the Epicenter) and the Inter Tribal Council of Arizona (ITCA). Randomization will occur regionally, at the site (schools and BGCs) level, to one of two conditions: IYG-AI/AN and a comparison condition. The comparison condition will consist of two web-based educational programs unrelated to sexual health. The IYG-AI/AN intervention will be compared against the comparison condition. The efficacy trial will continue for 16 months into year 4 (2013).

The primary hypothesis to be tested is: (1) youth who receive the IYG-AI/AN intervention will delay sexual activity relative to those who receive the comparison condition. The major dependent variable is the proportion of AI/AN youth initiating sexual activity (vaginal, oral, or anal sex). Secondary hypotheses will examine the effect of the intervention on specific types of sex (e.g., vaginal, oral, anal) and psychosocial variables such as youth intentions, knowledge, self-efficacy, attitudes, and perceived norms related to sexual risk-taking behavior. Secondary hypotheses will also examine the effect of the intervention on the proportion of AI/AN youth who are sexually active, occurrences of unprotected sexual intercourse and the number of sexual partners among these AI/AN youth.

ELIGIBILITY:
Inclusion Criteria:

* American Indian or Alaska Native descent and/or tribal affiliation
* Youth ages 12-14 attending regular classes in regional middle schools or youth attending after-school programs and/or Boys and Girls Clubs
* English-speaking

Exclusion Criteria:

* Youth who are not of American Indian or Alaska Native descent
* Any physical or mental condition that would inhibit the ability to complete surveys and use computer programs, such as cognitive impairment, motor disorders (e.g. quadriplegia), learning difficulties or psychiatric/behavioral problems (e.g. autism, attention deficit disorder)
* Students will be informed that the surveys and intervention materials will only be available in English and will be asked to consider their comfort level with participating in the study

Ages: 12 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 574 (Actual)
Dates: Start 2010-09; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Delay onset of sexual activity | baseline
  delay onset of vaginal, oral or anal sex
Delay onset of sexual activity | 5-months
  delay onset of vaginal, oral or anal sex
Delay onset of sexual activity | 16-months
  delay onset of vaginal, oral or anal sex

SECONDARY OUTCOMES:
Reduce alcohol/drug use | baseline
Reduce instances of sexual activity | baseline
Decrease the number of sexual partners | baseline
Condom use during sexual activity | baseline
Contraceptive use while sexually active | baseline
Prevalence of sexually transmitted infections | baseline
Increase sexual knowledge | baseline
Changes in sexual beliefs | baseline
Changes in attitudes toward sexual activity | baseline
Changes in perception of sexual beliefs among peers | baseline
Increased self-efficacy for refusal skills | baseline
Increased self-efficacy for condom use | baseline
Increased avoidance of risky situations | baseline
Changes in perceived norms about sexual activity | baseline
Changes in reasons for or against having sex | baseline
Changes in intentions to have/abstain from sex | baseline
Reduce alcohol/drug use | 5-months
Reduce alcohol/drug use | 16-months
Reduce instances of sexual activity | 5-months
Reduce instances of sexual activity | 16-months
Decrease the number of sexual partners | 5-months
Decrease the number of sexual partners | 16-months
Condom use during sexual activity | 5-months
Condom use during sexual activity | 16-months
Contraceptive use while sexually active | 5-months
Prevalence of sexually transmitted infections | 5-months
Prevalence of sexually transmitted infections | 16-months
Increase sexual knowledge | 5-months
Increase sexual knowledge | 16-months
Changes in sexual beliefs | 5-months
Changes in sexual beliefs | 16-months
Changes in attitudes toward sexual activity | 5-months
Changes in attitudes toward sexual activity | 16-months
Changes in perception of sexual beliefs among peers | 5-months
Changes in perception of sexual beliefs among peers | 16-months
Increased self-efficacy for refusal skills | 5-months
Increased self-efficacy for refusal skills | 16-months
Increased self-efficacy for condom use | 5-months
Increased self-efficacy for condom use | 16-months
Increased avoidance of risky situations | 5-months
Increased avoidance of risky situations | 16-months
Changes in perceived norms about sexual activity | 5-months
Changes in perceived norms about sexual activity | 16-months
Changes in reasons for or against having sex | 5-months
Changes in reasons for or against having sex | 16-months
Changes in intentions to have/abstain from sex | 5-months
Changes in intentions to have/abstain from sex | 16-months

CONTACTS AND LOCATIONS:
Overall Officials: Ross Shegog, PhD, Principal Investigator — The University of Texas Health Science Center, Houston; Christine Markham, PhD, Principal Investigator — The University of Texas Health Science Center, Houston; Melissa Peskin, DrPH, Principal Investigator — The University of Texas Health Science Center, Houston; Cornelia Jessen, MA, Principal Investigator — Alaska Native Tribal Health Consortium; Stephanie Craig-Rushing, MPH, PhD, Principal Investigator — Northwest Portland Area Indian Health Board; Gwenda Gorman, Principal Investigator — Inter Tribal Council of Arizona, Inc.; Scott Tulloch, Principal Investigator — Indian Health Service (IHS)
Locations (4):
- United States (4):
  - Alaska Native Tribal Health Consortium, Anchorage, Alaska
  - Inter Tribal Council of Arizona, Inc., Phoenix, Arizona
  - Northwest Portland Area Indian Health Board, Portland, Oregon
  - University of Texas Health Science Center, Houston, Houston, Texas

REFERENCES:
- [Derived] Markham CM, Craig Rushing S, Jessen C, Gorman G, Torres J, Lambert WE, Prokhorov AV, Miller L, Allums-Featherston K, Addy RC, Peskin MF, Shegog R. Internet-Based Delivery of Evidence-Based Health Promotion Programs Among American Indian and Alaska Native Youth: A Case Study. JMIR Res Protoc. 2016 Nov 21;5(4):e225. doi: 10.2196/resprot.6017. PMID 27872037